CLINICAL TRIAL: NCT03920462
Title: Evaluation of a Physical Activity Programme Using an Intelligent Electric Bike for Health in Healthy Volunteers.
Brief Title: Evaluation of a Physical Activity Programme Using an Intelligent Electric Bike for Health in Healthy Volunteers (PROTOVELIS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratoire TIMC-IMAG (Other)
Collaborators: TIMC-IMAG (Other); Floralis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-A00997-50
Record Dates: First submitted 2019-04-12; First posted 2019-04-19 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Physical Activity; Intelligent Electric Bike for Health; Connected Vest
Keywords: Physical Activity; Connected bike; Connected vest; Rehabilitation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: All volunteers realise a programme of 6 excursions with intelligent electric bike for health and connected vests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Programme of intelligent electric bike for health (single arm) (Other): All volunteers will realise the programme of intelligent electric bike for health with connected vests.
  Interventions: Device: Programme of intelligent electric bike for health

INTERVENTIONS:
Device: Programme of intelligent electric bike for health — It is a programme of 6 excursions with an intelligent electric bike for health and connected vests during 1 month (two excursions per week according the weather)

SUMMARY:
The walk and bike practice are two physical activities the most cited for benefits of physical activity thanks to their progressive and soft characters adapted to patients suffering from chronic diseases (diabetes, obesity, cancer...) with muscular deficit cardio-respiratory.

However, cycling may, depending on the natural land, imply efforts and articular-muscular-tendon pressions more important particularly in hilly natural land.

Moreover, lots of physical and physiological barriers oppose to the bike practice in the population of patients with chronic diseases. The electric bike can be useful.

This electric bike will be powerful but safe, totally programmable to adapt to patients, slope, rehabilitation objectives but very easy to use.

From medicine, it is necessary to ensure a moderate and regular effort regarding patients.

To do this, it is necessary to individualize adjustments of electric bike to have a progressive rehabilitation program and a progressive load force.

It needs to dispose monitoring and evaluation tools in real situations outside (lots of physiological and technical sensors). The intelligent electric bike for health proposes to be in accordance to this specifications.

DETAILED DESCRIPTION:
The investigators propose to validate the technical and organizational feasibility of workshops using the intelligent electric bike for health with different devices such as two connected vests (non-invasive) measuring on the one hand the cardiological and respiratory parameters (connected vest named : Etisens) and the other hand the kinetic energy of movement (connected vest named : Optimove).

The development of this ambulatory physiology platform and the engine brake create perspectives for an outdoor rehabilitation tool that for example could stimulate, on an altitude free-excursion, a mountain pass of Alpes doing the link of health, sport and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to ride a bike
* Volunteer without a contraindication to moderate physical activity or cycling (acute coronary artery disease less than 2 years old, musculoskeletal problem of the spine or lower limbs incompatible with cycling).
* weight < 125 kg
* volunteer available for an intervention of 2-3 hours twice a week during 1 month.

Exclusion Criteria:

* Person deprived of liberty or legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of intelligent electric bike for health programme validated evaluated by the questionnaire "evaluation of the programme of intelligent electric bike for health - volunteer". | 1 month
  Score of questionnaire "evaluation of the programme of intelligent electric bike for health - volunteer". A negative value is defined by a value less than 5 and a positive value is defined by a value greater than 5.

SECONDARY OUTCOMES:
Percentage of excursions validated evaluated by the questionnaire "excursion evaluation - volunteer". | 1st week, 2nd week, 3rd week and 4th week.
  Score of questionnaire "excursion evaluation - volunteer" for each excursion. A negative value is defined by a value less than 5 and a positive value is defined by a value greater than 5.
Percentage of specific characteristics validated for each excursion evaluated by the questionnaire "excursion evaluation - volunteer". | 1st week, 2nd week, 3rd week and 4th week.
  Score of items 1, 2 and 3 of questionnaire "excursion evaluation - volunteer" for each excursion.
  For item 1 and 2 ; a negative value is defined by a value less than 4 and greater than 6, and a positive value by a value between 4 and 6.
  For item 3 ; a negative value is defined by a value less than 5 and a positive value is defined by a value greater than 5.
Percentage of general characteristics validated for each excursion evaluated by the questionnaire named "excursion evaluation - volunteer". | 1st week, 2nd week, 3rd week and 4th week.
  Score of items 1, 2, 3, 4 and 5 of questionnaire "excursion evaluation - volunteer" for each excursion.
  A negative value is defined by a value less than 5 and a positive value is defined by a value greater than 5.
Percentage of excursions validated evaluated by the questionnaire "excursion evaluation - supervising staff". | 1st week, 2nd week, 3rd week and 4th week.
  Score of questionnaire "excursion evaluation - supervising staff" for each excursion. A negative value is defined by a value less than 5 and a positive value is defined by a value greater than 5.
Percentage of specific characteristics validated for each excursion evaluated by the questionnaire "excursion evaluation - supervising staff". | 1st week, 2nd week, 3rd week and 4th week.
  Score of items 1,2 and 3 of questionnaire "excursion evaluation - supervising staff" for each excursion. A negative value is defined by a value less than 5 and a positive value is defined by a value greater than 5.
Percentage of general characteristics validated for each excursion evaluated by the questionnaire "excursion evaluation - supervising staff". | 1st week, 2nd week, 3rd week and 4th week.
  Score of items 1, 2, 3, 4 and 5 of questionnaire "excursion evaluation - supervising staff" for each excursion.
  A negative value is defined by a value less than 5 and a positive value is defined by a value greater than 5.
Percentage of programme validated evaluated by the questionnaire "evaluation of the programme of intelligent electric bike for health - supervising staff". | 1 month
  Score of questionnaire "evaluation of the programme of intelligent electric bike for health - supervising staff". A negative value is defined by a value less than 5 and a positive value is defined by a value greater than 5.
Percentage of data stored by the intelligent electric bike for health. | 1st week, 2nd week, 3rd week and 4th week.
  The validation of records is defined when 90% of data is saved.
Percentage of data stored by the connected vest Etisense. | 1st week, 2nd week, 3rd week and 4th week.
  The validation of records is defined when 90% of data is saved, all sensors are functional and data are relevant.
Comparison between data stored by the connected vest Etisense and the intelligent electric bike for health. | 1st week, 2nd week, 3rd week and 4th week.
  Respiratory rate of the connected vest Etisense and the intelligent electric bike for health are compared.
Percentage of data stored by the connected vest Optimove. | 1st week, 2nd week, 3rd week and 4th week.
  The validation of records is defined when 90% of data is saved.
Compare data stored by the connected vest Optimove during two excursions with adjustments different of the intelligent electric bike for health. | 1st week, 2nd week, 3rd week and 4th week.
  Data of the connected vest Optimove and the intelligent electric bike for health are compared.
Comparison between theoretical speed limit and real speed observed. | 1 month
  Speed recorded by the intelligent electric bike for health (real speed observed) and theoretical speed (programmed speed) are compared.
Capacity of the intelligent electric bike for health to offer entrainment capacities for a high-level athlete. | 1 month
  Description of features of the intelligent electric bike for health for entrainment of high-level athlete.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-luc BOSSON, Principal Investigator — TIMC-IMAG
Locations (1):
- BOSSON Jean-Luc, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pavey TG, Anokye N, Taylor AH, Trueman P, Moxham T, Fox KR, Hillsdon M, Green C, Campbell JL, Foster C, Mutrie N, Searle J, Taylor RS. The clinical effectiveness and cost-effectiveness of exercise referral schemes: a systematic review and economic evaluation. Health Technol Assess. 2011 Dec;15(44):i-xii, 1-254. doi: 10.3310/hta15440. PMID 22182828
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A; American College of Sports Medicine; American Heart Association. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Circulation. 2007 Aug 28;116(9):1081-93. doi: 10.1161/CIRCULATIONAHA.107.185649. Epub 2007 Aug 1. PMID 17671237
- [Background] Peterman JE, Morris KL, Kram R, Byrnes WC. Pedelecs as a physically active transportation mode. Eur J Appl Physiol. 2016 Aug;116(8):1565-73. doi: 10.1007/s00421-016-3408-9. Epub 2016 Jun 14. PMID 27299435
- [Background] Gojanovic B, Welker J, Iglesias K, Daucourt C, Gremion G. Electric bicycles as a new active transportation modality to promote health. Med Sci Sports Exerc. 2011 Nov;43(11):2204-10. doi: 10.1249/MSS.0b013e31821cbdc8. PMID 22005715
- [Background] Welker J, Cornuz J, Gojanovic B. [Electrically assisted bicycles: health enhancement or "green" gadget?]. Rev Med Suisse. 2012 Jul 25;8(349):1513-7. French. PMID 22913003
- See also: Des Asters R. The impact evaluation on the health, promotion of electric bike. 2006 — http://www.impactsante.ch/pdf/EIS_VAE_2006.pdf
- See also: Gretchen Reynolds. The Surprising Health Benefits of an Electric Bike. 2016 — http://well.blogs.nytimes.com/2016/07/06/the-surprising-health-benefits-of-an-electric-bike-2/?smid=tw-nytimes&smtyp=cur&_r=1